CLINICAL TRIAL: NCT07213596
Title: Development of Virtual Reality Treatment Technology to Treat Trauma Related to COVID-19 Infection
Brief Title: Virtual Reality Treatment for Trauma Related to COVID-19 Infection
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Ji Sun Kim, Professor, Soonchunhyang University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHCA IRB 2022-08-032-033; RS-2022-KH125605 (Other Grant/Funding Number: the Ministry of Health and Welfare, Republic of Korea)
Record Dates: First submitted 2025-10-01; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: PTSD; PTSD Symptoms
Keywords: VR exposure; PTSD symptoms; covid 19
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; COVID-19 | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthcare workers with VR Exposure Therapy (Experimental): Healthcare workers with VR Exposure Therapy with 5 sessions weekly
  Interventions: Behavioral: VR Exposure Therapy
- COVID-19 survivors with VR Exposure Therapy (Experimental): general population with VR Exposure Therapy with 5 sessions weekly
  Interventions: Behavioral: VR Exposure Therapy
- Healthcare workers with CBT (Active Comparator): Healthcare workers with CBT with weekly 5 sessions
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- COVID-19 survivor with Supportive Therapy/TAU (Active Comparator): individual recovered from COVID-19 with Supportive Therapy/TAU
  Interventions: Behavioral: Supportive Psychotherapy

INTERVENTIONS:
Behavioral: VR Exposure Therapy — Virtual Reality Exposure Therapy (VRET) is a form of psychotherapy that uses immersive virtual environments to simulate trauma-related stimuli in a controlled and safe setting, allowing individuals to gradually confront and process distressing memories or triggers.
  VRET is grounded in prolonged exposure (PE) therapy, a well-established treatment for PTSD and anxiety disorders.
  In this study, VRET is delivered in 5 weekly sessions, each lasting approximately 50 minutes, using a customized VR system.
  Sessions are tailored based on participant group (e.g., COVID-19 survivor vs. healthcare worker).
  Each session includes psychoeducation, exposure to individualized trauma-related virtual scenes, and guided emotional processing.
  The system incorporates eye-tracking, breathing exercises, and real-time subjective distress scaling (SUDs) to monitor engagement and safety.
  Arms: COVID-19 survivors with VR Exposure Therapy; Healthcare workers with VR Exposure Therapy
Behavioral: Cognitive Behavioral Therapy (CBT) — Face-to-face CBT with exposure elements, targeting trauma-related symptoms. Administered in 5 weekly sessions.
  Arms: Healthcare workers with CBT
Behavioral: Supportive Psychotherapy — Therapist-led supportive therapy (TAU), focusing on empathy, validation, and emotional support without structured exposure.
  Arms: COVID-19 survivor with Supportive Therapy/TAU

SUMMARY:
This clinical trial aims to develop and evaluate the effectiveness of virtual reality (VR)-based exposure therapy for trauma symptoms related to COVID-19 infection. The intervention targets healthcare workers and individuals from the general population who experienced pandemic-related psychological distress. The study assesses psychological and physiological outcomes, including PTSD, anxiety, depression, HRV, and EEG biomarkers.

DETAILED DESCRIPTION:
The project involves a two-phase clinical study. In Phase 1, VR exposure therapy content is developed based on trauma management theory and tailored to specific participant groups (e.g., COVID-19 survivors, healthcare workers). In Phase 2, randomized controlled trials will compare VR treatment with standard therapy approaches (CBT, supportive therapy) across two populations:

Healthcare workers involved in the care of COVID-19 patients Members of the general public affected by social disaster-related psychological distress

Participants will undergo 5 weekly sessions of VR exposure therapy. Pre- and post-intervention assessments will include standardized psychiatric scales (e.g., PHQ-9, PCL-5), HRV, and EEG measurements. The trial aims to validate the efficacy and safety of customized VR therapy protocols and identify relevant biomarkers for treatment prediction.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64, healthy population who survived from COVID-19 (COVID survivors) or Healthcare Workers with PCL-5 ≥10, GAD-7/PHQ-9 ≥10

Exclusion Criteria:

* Pregnancy, neurological disorders, severe medical conditions

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD symptoms | baseline, week 5, 3-mo follow-up
  Change in PTSD symptoms (PCL-5/CAPS-5) at baseline, week 5, 3-mo follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ji Sun Kim, MD, PhD, Principal Investigator — Soonchunhyang University Hospital

IPD SHARING:
Plan to Share IPD: No
No. Individual participant data (IPD) will not be shared due to confidentiality concerns and regulatory restrictions.